CLINICAL TRIAL: NCT07223398
Title: STOP (Shared Decision Making to Treat Or Prevent) HIV in Justice Populations
Brief Title: Shared Decision Making to Treat Or Prevent (STOP) HIV in Justice Populations (R33)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000037052_a; 4R33DA060625-02 (NIH)
Record Dates: First submitted 2025-10-30; First posted 2025-10-31 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders | interventions — Patient Freedom of Choice Laws

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Patient Navigation (PN) (Active Comparator): PNs are "near-peer" professionals who have shared lived experiences with participants and help them overcome barriers to accessing and engaging in quality care. PNs are trained and linked to PrEP/ART and SUD services. This manualized PN approach provides a complete assessment of participant needs, goal setting, and help with appointment scheduling.
  Interventions: Behavioral: Standard PN
- PN + Patient Choice (PC) (PN+PC) (Experimental): PNs working in the PN + PC arm will be trained to engage participants in selecting from a menu of service options in their community. This menu of SUD and HIV prevention and treatment service delivery options will be created through bolstering and working with our Community Advisory Boards (CAB). PNs will also be trained to discuss sexual and substance use history with participants in order to provide education and motivation towards starting PrEP/ART and SUD treatment.
  Interventions: Behavioral: Standard PN; Behavioral: Patient Choice

INTERVENTIONS:
Behavioral: Standard PN — Standard of care
Behavioral: Patient Choice — Participants can select from a menu of options including brick and mortar services, Mobile Health Unit (MHU) or telehealth services.
  Arms: PN + Patient Choice (PC) (PN+PC)

SUMMARY:
This study seeks to compare the effectiveness of two Patient Navigation models of care to evaluate the proportion who initiate PrEP/ART and substance use/substance use disorder (SU/SUD) treatment. A standardized Patient Navigation (PN) arm will be compared with a shared decision-making model in the form of Patient Choice (PC) through the offer of a menu of existing community-based health service delivery options. This design will offer providers, correctional and public health authorities, payers and policy makers' timely and relevant data to assess the effectiveness of Patient Navigation and Patient Choice models of care as potentially useful re-entry and relapse prevention treatment options.

DETAILED DESCRIPTION:
This study will be done in two phases. Aim 1, the R61 portion of the project will be a Pilot Study, and Aim 2, the R33 portion of the project will be a Randomized Controlled Trail informed by the pilot.

The focus of this registration is Aim 2, the randomized controlled trial. The Aim 1 (R61) portion is registered with NCT06439329. In Aim 2 (R33), investigators will evaluate standard PN compared to PN+PC on participant outcomes, implementation outcomes and costs associated with implementing the study.

ELIGIBILITY:
Inclusion Criteria:

* able to provide written informed consent in English or Spanish;
* living in the community of Western, CT, Dallas and Tarrant Counties in TX and Madison County, KY (potential for Fayette county as well);
* Those with current justice involvement (with in the past 6 months) (e.g., prison, jail, community supervision);
* willing to have HIV testing to determine negative or positive status;
* persons with HIV who report not currently taking ART in past 6 months OR persons who test negative for HIV who report not taking PrEP that meet CDC PrEP eligibility criteria in past 6 months, including (i) condomless sexual intercourse; and/or (ii) sharing IDU equipment with HIV positive or unknown status partner; and/or (iii) bacterial STI and;
* Having a history of opioid and/or stimulant use in the last 6 months within the community.

Exclusion Criteria:

* severe medical or psychiatric disability making participation unsafe;
* unable to provide consent.
* persons self-reporting pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who initiate or re-initiate PrEP | 6 months
  Percentage of participants not living with HIV who initiate or re-initiate PrEP within the 6-month intervention period by self report
Percentage of participants who initiate or re-initiate ART | 6 months
  Percentage of participants living with HIV who initiate or re-initiate ART within the 6-month intervention period by self report

SECONDARY OUTCOMES:
Percentage of participants that adhere to PrEP | 6 and 12 months
  Percentage of participants that adhere to PrEP
Percentage of participants retaining on PrEP | 6 and 12 months
  Percentage of participants retaining on PrEP
HIV incidence | 6 and 12 months
  HIV incidence [binary] for those testing negative using rapid point of care (POC) test over time
Percentage of participants that adhere to ART | 6 and 12 months
  Percentage of participants that adhere to ART
ART retention | 6 and 12 months
  For persons living with HIV (PLH), ART retention [binary]
Substance use treatment | 6 and 12 months
  Percentage of participants engaged in substance use disorder (SUD) treatment
HIV viral suppression | 6 months
  For PLH, HIV viral suppression, for those with HIV at time of randomization: the percent who maintain or achieve HIV viral load < 200 copies/mL at 6 months
Retention in HIV PrEP/ART | 6 months
  Retention in HIV PrEP/ART care [binary]: defined as attending 2 or more visits in 6-months
Number of Participants Who Had Any Needle Sharing Activity to Assess HIV Risk Behavior | 6 and 12 months
  Number of Participants Who Had Any Needle Sharing Activity
Number of Participants Who Had Sex Without a Condom to assess HIV Risk Behavior | 6 and 12 months
  Number of Participants Who Had Vaginal or Anal Sex Without a Condom
Days of using opioids | 6 and 12 months
  Measured by Timeline Followback, which assesses self-reported alcohol and other drug use including opioid use
Number of participants with with overdose events | 6 and 12 months
  Number of participants with non-fatal and fatal overdose events
Percentage of participants with retention in SUD treatment | 6 and 12 months
  Retention in SUD treatment including but not exclusive to Medication for Opioid Use Disorder (MOUD) for Opioid Use Disorder (OUD)
Quality of Life assessed using PROMIS-PROPr | 6 and 12 months
  PROMIS-PROPr assesses general societal health. Total summary score ranges from -0.022, worse than dead, to 1, perfect health.
Change in Depression assessed using Patient Health Questionnaire-9 (PHQ-9) | 6 and 12 months
  Depression will be assessed using the PHQ-9. PHQ-9 is a 9-item validated questionnaire used to screen for depression with a range of scores from 0-45. A cumulative score of ≥10 is considered positive with lower scores indicating no or mild anxiety.
Recidivism: Reasons | 6 and 12 months
  Number of participants per reason for arrest/ incarceration/return-to-custody
Recidivism: Mean days in custody/incarcerated | 6 and 12 months
  Mean days in custody/incarcerated
Recidivism: Mean days to return | 6 and 12 months
  Mean days to return to custody/incarcerated
HIV and SU Stigma assessed using Substance Use Stigma Mechanisms Scale (SU-SMS) | 6 and 12 months
  Mean score for Enacted (6 items), Anticipated (6 items), and Internalized (6 items) scales. Each scale is scored 1-5, with higher scores indicating greater endorsement of substance use stigma
Percentage of participants diagnosed with SUD | Baseline and 12 months
  Percentage of participants diagnosed with SUD using DSM-5

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Springer, MD, Principal Investigator — Yale University
Locations (4):
- United States (4):
  - Yale School of Medicine, New Haven, Connecticut
  - College of Medicine at the University of Kentucky, Lexington, Kentucky
  - University of Texas Southwestern Medical Center (UTSW), Dallas, Texas
  - Texas Christian University's (TCU) School of Medicine, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: No